CLINICAL TRIAL: NCT01618643
Title: Acetowhitening Time as a Novel Objective Tool for the Diagnosis of High Risk Neoplasia in Barrett's Oesophagus
Brief Title: Aceto-whitening in the Assessment of Gastrointestinal Neoplasia
Status: Completed | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Collaborators: University of Portsmouth (Other)
Responsible Party: Sponsor
Other Study IDs: PHT/2010/25
Record Dates: First submitted 2012-06-11; First posted 2012-06-13 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Barrett Esophagus; Barrett Metaplasia; Barrett Oesophagitis With Dysplasia; Barrett Adenocarcinoma
Keywords: Barrett's; High grade dysplasia; HGD; IMC; Intramucosal cancer; Acetic acid; Chromoendoscopy
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Only pathology retained is for NHS purposes only. No separate tissue retained for the study
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Acetic acid chromoendoscopy: * Patients with known Barrett's metaplasia under surveillance
  * Patients with Barrett's metaplasia who had undergone endoscopic treatment for neoplasia previously and were under surveillance for metachronous neoplasia
  * Patients suspected of neoplasia referred for endoscopic mucosal resection or other targeted endoscopic treatment of the lesion
  Interventions: Procedure: Acetic acid chromoendoscopy

INTERVENTIONS:
Procedure: Acetic acid chromoendoscopy — Prospective observational pilot study.
  We would examine patients with Barrett's epithelium that is either healthy or has suspected areas of neoplasia. We will apply acetic acid spray to areas of healthy Barrett's metaplasia and time how long it takes for the aceto whitening to disappear. We will repeat this in cases referred with SM invasive cancer, intramucosal cancer, suspected high grade dysplasia and possible low grade dysplasia. We will record how long it takes for the acetowhitening to disappear. We will biopsy these areas to confirm the diagnosis.
  We will correlate the histology to the aceto-whitening time to see if there is a correlation between the degree of neoplasia and the aceto-whitening time after acetic acid dye spray.

SUMMARY:
Acetic acid chromoendoscopy is an established standard technique used to detect dysplasia within the gastrointestinal tract. Acetic acid spray helps to identify neoplasia by highlighting the surface pattern, highlighting the vascular pattern and by a process known as the aceto-whitening reaction, where tissues take acetic acid and turn white for a brief period and then slowly revert back to a normal colour. The neoplastic surface and vascular pattern are all very well described, and have played a big role in the recognition of early cancer. The aceto-whitening reaction is well described but the differential in timing between neoplastic and non-neoplastic areas is not well understood.

The investigators aim to establish the differential in the timing of the disappearance of the aceto-whitening reaction between healthy tissue, dysplastic tissue, intramucosal cancer and invasive cancer after acetic acid dye spray in the oesophagus and colon. By understanding this better, the investigators may be able to predict with greater accuracy whether a highlighted abnormal area is cancer or high grade dysplasia, or whether it is low grade dysplasia or inflammation, which has significant prognostic implications for the patient.

The investigators hypothesize that the differential in the timing of the disappearance of the aceto-whitening reaction between normal and abnormal tissue could help in the detection of gastrointestinal neoplasia.

DETAILED DESCRIPTION:
This is a prospective pilot study. It is standard practice within our unit to use acetic acid for the detection of neoplasia. No patient would receive any additional intervention that would not normally be performed.

We will record the surface and vascular patterns before and after acetic acid spray. As usual we will then apply acetic acid spray to the Barrett's epithelium and time how long it takes for the aceto whitening to disappear. It is the timing of the disappearance that is the key study intervention. We will biopsy these areas to confirm the diagnosis. Again this is standard practice and no patient will be denied an intervention that is normally performed, and no extra interventions will be performed over and above the standard clinical practice.

We will correlate the histology to the aceto-whitening disappearance time to identify a threshold time which can serve as a cut off between neoplastic and non-neoplastic tissue.

We hypothesise that the aceto-whitening reaction lasts much longer in the normal epithelium of Barrett's oesophagus and colon. This reaction will be much shorter in areas with abnormal pathology like dysplasia or cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known Barrett's metaplasia under surveillance
* Patients with Barrett's metaplasia who had undergone endoscopic treatment for neoplasia previously and were under surveillance for metachronous neoplasia
* Patients suspected of neoplasia referred for endoscopic mucosal resection or other targeted endoscopic treatment of the lesion

Exclusion Criteria:

* Oesophagitis
* Contact bleeding
* Acute mucosal trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surveillance for Barrett's oesophagus
Sampling Method: Non-Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2010-11-23 (Actual); Primary Completion 2011-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Timing of disappearance of aceto-whitening for Barrett's metaplasia, HGD and cancer | 18 months
  To quantify the differential in the timing of the disappearance of the aceto-whitening reaction between metaplastic tissue, dysplastic tissue and invasive cancer after acetic acid dye spray in the oesophagus and colon.

SECONDARY OUTCOMES:
To differentiate mucosal neoplasia from invasive cancer | 24 months
  To differentiate high grade displasia and intramucosal cancer from invasive cancer using the aceto-whitening timing

CONTACTS AND LOCATIONS:
Overall Officials: Pradeep Bhandari, MD, FRCP, Principal Investigator — Portsmouth Hospitals NHS Trust
Locations (1):
- Portsmouth Hospitals NHS trust, Portsmouth, Hampshire, United Kingdom